CLINICAL TRIAL: NCT02122536
Title: Split-Face, Double-blind, Single Center, Prospective Study Comparing OnabotulinumtoxinA to IncobotulinumtoxinA
Brief Title: Split-Face Prospective Study Comparing Botox to Xeomin for the Treatment of Facial Wrinkles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: YMD Eye and Face (Other)
Responsible Party: Principal Investigator, Ruth Hill Yeilding, MD, YMD Eye and Face
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 318060-3
Record Dates: First submitted 2013-10-30; First posted 2014-04-24 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Facial Wrinkles
MeSH Terms: interventions — incobotulinumtoxinA; Random Allocation; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Xeomin right side; Xeomin to left side of face (Active Comparator): Patients were randomized as to which side of the face was treated with Xeomin.
  Interventions: Drug: Xeomin to right side of face in half of the subjects; Xeomin to left side of face in the other half of subjects
- Botox right side; Botox to left side (Active Comparator): Patients were randomized as to which side of the face was treated with Botox.
  Interventions: Drug: Botox to right side of face in half of the subjects (randomized); Botox to the left side of the face in the other half of subjects

INTERVENTIONS:
Drug: Xeomin to right side of face in half of the subjects; Xeomin to left side of face in the other half of subjects — Subjects were randomized to which side of the face would be treated with Xeomin.
  Other Names: incobotulinumtoxinA (Xeomin)
  Arms: Xeomin right side; Xeomin to left side of face
Drug: Botox to right side of face in half of the subjects (randomized); Botox to the left side of the face in the other half of subjects — Subjects were randomized to which side of the upper face would be treated with Botox
  Other Names: onabotulinumtoxinA (Botox)
  Arms: Botox right side; Botox to left side

SUMMARY:
The aim of this prospective, randomized, double-blind, intraindividual split face study will be to compare onabotulinumtoxinA to incobotulinumtoxinA for the correction of facial wrinkles using a 1:1 dose ratio.

DETAILED DESCRIPTION:
Patients will be randomized to which side of the face will be injected with onabotulinumtoxinA and incobotulinumtoxinA. A total dose of 22.5 units of onabotulinumtoxinA and 22.5 units of incobotulinumtoxinA will be administered at baseline to the respected side of the face. One vial (100 MU) of BoNTA will be reconstituted with 2.0 mL of 0.9% sterile saline solution. Similarly, one vial (100 MU) of BTXCo will be reconstituted with 2.0 mL of 0.9% sterile saline solution. 2.5 units of the respective neurotoxin will be administered to three sites in the crow's feet area on each side (7.5 units total for one side), 2.5 units to two locations of the forehead on each side (5 units total for one side), and 5.0 units to two locations in the glabella on each side(10 units total for one side). The duration of the study will be 4 months. The followup visits after the initial injections will be at 3 days, 2 weeks, 3 months, and 4 months after the initial treatment. At each of these visits, standardized digital photographs of the treated facial area will be taken. Both static and dynamic photos will be taken of each region. At the conclusion of the study, three independent raters will individually perform blind assessments of the photographs according to the Validated Assessment Scaled for the Upper Face published by Flynn et al 2012.

ELIGIBILITY:
Inclusion Criteria:

* males and females age 18 or older.

Exclusion Criteria:

* Previous treatment with a neuromodulator in the last 6 months
* previous brow lift
* currently pregnant or breastfeeding
* a history of neurological disease or deficit
* an active facial skin infection
* an allergy to neuromodulators

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-07; Primary Completion 2012-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in Wrinkles Score | Preinjection assessment; assessment at 3 days, 2 weeks, 3 months, 4 months post-injection
  Objective assessment of change in wrinkles score pre and post injection of the crow's feet, glabella, and forehead using the "Validated Assessment Scaled for the Upper Face" published by Flynn et al. 2012. At the end of the study the delta wrinkle score from pre-injection to each followup assessment for each area will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth H Yeilding, MD, Principal Investigator — YMD Eye & Face
Locations (1):
- Center for Sight, Sarasota, Florida, United States

REFERENCES:
- [Background] Flynn TC, Carruthers A, Carruthers J, Geister TL, Gortelmeyer R, Hardas B, Himmrich S, Kerscher M, de Maio M, Mohrmann C, Narins RS, Pooth R, Rzany B, Sattler G, Buchner L, Benter U, Fey C, Jones D. Validated assessment scales for the upper face. Dermatol Surg. 2012 Feb;38(2 Spec No.):309-19. doi: 10.1111/j.1524-4725.2011.02248.x. PMID 22316187
- [Derived] Yeilding RH, Fezza JP. A Prospective, Split-Face, Randomized, Double-Blind Study Comparing OnabotulinumtoxinA to IncobotulinumtoxinA for Upper Face Wrinkles. Plast Reconstr Surg. 2015 May;135(5):1328-1335. doi: 10.1097/PRS.0000000000001255. PMID 25919246